CLINICAL TRIAL: NCT00513539
Title: Porfimer Sodium Photodynamic Therapy Plus Stenting Versus Stenting Alone in Patients With Advanced or Metastatic Cholangiocarcinomas and Other Biliary Tract Tumours: a Multicentre, Randomised, Phase Lll Study
Brief Title: Biliary Stenting With or Without Photodynamic Therapy in Treating Patients With Locally Advanced, Recurrent, or Metastatic Cholangiocarcinoma or Other Biliary Tract Tumors That Cannot Be Removed by Surgery
Acronym: Photostent-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000558540; CRUK-PHOTOSTENT-02; EU-20740; EUDRACT-2005-001173-96; ISRCTN87712758; CTA-20363/0207/001-0001
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer
Keywords: unresectable gallbladder cancer; recurrent gallbladder cancer; metastatic gallbladder cancer; cholangiocarcinoma of the gallbladder; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; metastatic extrahepatic bile duct cancer; cholangiocarcinoma of the extrahepatic bile duct
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Biliary Stenting alone
  Interventions: Procedure: biliary stenting
- Arm B (Experimental): Photodynamic Therapy plus biliary stenting
  Interventions: Drug: porfimer sodium; Procedure: biliary stenting

INTERVENTIONS:
Drug: porfimer sodium
  Arms: Arm B
Procedure: biliary stenting

SUMMARY:
RATIONALE: Biliary stenting is the placement of a tube in the bile ducts to keep a blocked area open. Photodynamic therapy uses a drug, such as porfimer sodium, that is absorbed by tumor cells. The drug becomes active when it is exposed to light. When the drug is active, tumor cells are killed. It is not yet known whether biliary stenting is more effective with or without photodynamic therapy in treating patients with biliary tract tumors.

PURPOSE: This randomized phase III trial is studying biliary stenting to see how well it works compared with biliary stenting and photodynamic therapy using porfimer sodium in treating patients with locally advanced, recurrent, or metastatic cholangiocarcinoma or other biliary tract tumors that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the efficacy, in terms of overall survival, of biliary stenting with vs without photodynamic therapy using porfimer sodium in advanced, recurrent, or metastatic biliary tract carcinoma.

Secondary

* To evaluate the two treatments arms with respect to progression-free survival, toxicity using NCI Common Toxicity Criteria (version 3.0), and quality of life.

OUTLINE: This is a multicenter study. Patients are stratified by participating center, primary site (gallbladder vs bile duct), disease stage (locally advanced vs metastatic), prior therapy (i.e., surgery, radiotherapy or chemotherapy) (yes vs no), performance score (0 vs 1 vs 2 vs 3), and prior treatment arm on UK chemotherapy trial ABC-02 (gemcitabine hydrochloride alone vs gemcitabine hydrochloride and cisplatin). Patients are randomized to 1 of 2 arms.

* Arm I: Patients undergo either endoscopic or percutaneous drainage and insertion of unilateral or bilateral plastic endoprostheses above the main strictures of the right and left hepatic bile ducts.
* Arm II: Patients undergo treatment as in arm I. Patients also receive porfimer sodium IV and then undergo laser activation 48 hours later.

After completion of study treatment, patients are followed every 3 months for at least 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histopathological/cytological diagnosis of nonresectable locally advanced, recurrent, or metastatic biliary tract carcinoma (intra- or extra-hepatic), or gallbladder carcinoma
* Adequate biliary drainage, with no evidence of active uncontrolled infection (patients on antibiotics are eligible)

Exclusion criteria:

* Porphyria
* No brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0, 1, 2, or 3
* Estimated life expectancy > 3 months
* Women of child-bearing potential should have a negative pregnancy test prior to study entry AND be using an adequate contraception method, which must be continued for 1 month after completion of treatment
* Not pregnant or nursing

Exclusion criteria:

* History of prior malignancy that will interfere with the response evaluation (exceptions include in-situ carcinoma of the cervix treated by cone-biopsy/resection, non-metastatic basal and/or squamous cell carcinomas of the skin, or any early stage (stage l) malignancy adequately resected for cure greater than 5 years previously)
* Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial
* Any psychiatric or other disorder likely to impact on informed consent

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Patients may have undergone a non-curative operation (i.e., R2 resection [with macroscopic residual disease] or palliative bypass surgery only) and fully recovered

  * Patients who have previously undergone curative surgery must have evidence of non-resectable disease relapse
* Patients may have received prior radiotherapy within the past 28 days (with or without radio-sensitizing low-dose chemotherapy) for localized disease and fully recovered

  * Must have clear evidence of disease progression prior to inclusion in this study
* Patients may have received prior chemotherapy within the past 28 days and fully recovered

  * Must have clear evidence of disease progression prior to inclusion in this study

Exclusion criteria:

* Previous treatment with curative intent for current disease in the last 12 weeks (i.e., prior resection, radical radiotherapy, or chemotherapy)
* Previous treatment with experimental therapy for current disease in the last 12 weeks
* No cytotoxic chemotherapy, radiotherapy, immunotherapy, hormonal therapy (excluding contraceptives and replacement steroids), or experimental medications will be permitted for the first four weeks of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | minimum follow up 3 years or until death

SECONDARY OUTCOMES:
Progression-free survival every 3 months | minimum follow up 3 years or until death
Toxicity as assessed by NCI CTC v. 3.0 | patients followed up for minimum of 3 years
Quality of life as assessed by EORTC QLQ 30 and PAN 26 at baseline and 1, 3, and 6 months after completion of study treatment | patients followed up for a minimum of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P. Pereira, MD, Study Chair — University College London Hospitals
Locations (4):
- United Kingdom (4):
  - Aintree University Hospital, Liverpool, England
  - University College Hospital, London, England
  - Queen's Medical Centre, Nottingham, England
  - Ninewells Hospital, Dundee, Scotland